CLINICAL TRIAL: NCT06190210
Title: The Impact of Perioperative Neurovascular Coupling on Outcome in Infants With Congenital Heart Disease.
Brief Title: Predictive Value of Neurovascular Coupling in Infants With COngenital Heart Disease
Acronym: NICO
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S68131
Record Dates: First submitted 2023-12-15; First posted 2024-01-05 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Congenital Heart Disease; Neurodevelopmental Disorders; Electroencephalography; Near-Infrared Spectroscopy; Biomarkers
Keywords: Congenital heart disease; Neurodevelopment; Neuromonitoring; Biomarkers; EEG; NIRS
MeSH Terms: conditions — Heart Defects, Congenital; Neurodevelopmental Disorders | interventions — Electroencephalography; Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — methylation patterns of neuronal cell-free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Congenital heart disease: Neonates with congenital heart disease necessitating treatment before the age of 6 months, either surgical or through cardiac catheterization
  Interventions: Diagnostic Test: electroencephalography; Diagnostic Test: Near-Infrared Spectroscopy; Diagnostic Test: neuronal cell-free DNA

INTERVENTIONS:
Diagnostic Test: electroencephalography — Pre-, per- and postoperative electroencephalography
  Other Names: EEG
Diagnostic Test: Near-Infrared Spectroscopy — Pre-, Per- and Postoperative near-infrared spectroscopy returning regional cerebral oxygen saturation
  Other Names: NIRS
Diagnostic Test: neuronal cell-free DNA — CfDNA which is characterized based on methylation patterns to determine the tissue of origin
  Other Names: cfDNA

SUMMARY:
Infants with congenital heart disease (CHD) are at increased risk for delayed neurodevelopment. Multiple etiological explanations have been proposed, as there seems to be a multifactorial interplay of both prenatal and perioperative factors. The main goal of this research project is to focus on peri-operative physiological risk factors in infants with CHD which impair functional brain maturation or elicit brain injury, and subsequently creating a risk model and guidelines for standardized developmental follow-up in this population.

PART 1: investigation of cerebral autoregulation and neurovascular coupling The homeostasis in cerebral blood supply regardless of perfusion pressure, is called Cerebral autoregulation (CAR). Neurovascular coupling (NVC) is the phenomenon in which blood supply increases as a result of increased brain activity in a specific area. At different times in the perioperative phase, these regulatory mechanisms will be estimated based on Electroencephalography (EEG) and Near Infrared Spectroscopy (NIRS), in addition to hemodynamic parameters.

PART 2: cell-free DNA (cfDNA) extraction. Non-invasive monitoring of neuronal degeneration can be performed using cfDNA extraction techniques. Serial measurements of neuronal cfDNA will be used to determine whether and when this neuronal damage has occurred.

PART 3: Prognosis and outcome. These risk factors, supplemented with demographic factors and medications administered, will be combined in an Artificial Intelligence-driven model, thus establishing a risk model for neurodevelopmental outcome. This model will be compared to the current standard-of-care, both structural imaging (ultrasound and MRI) and a clinical developmental assessment at 9 and 24 months of age (Bayley Scales of Infant Development-III).

ELIGIBILITY:
Inclusion Criteria:

* CHD warranting a first percutaneous or surgical intervention in the first 6 months, including but not limited to transposition of the great arteries (TGA), univentricular heart (UVH), Tetralogy of Fallot (TOF), coarctation of the aorta (CoA), total abnormal pulmonary venous drainage (TAPVU), Common arterial trunc (TA), large patent ductus arteriosus (PDA) or VSD and AVSD for which treatment is necessary within the first 6 months of life.
* Treatment provided at the University Hospitals Leuven.

Exclusion Criteria:

* Syndromes or proven genetic conditions which are associated with neurological impairment
* CHD warranting treatment after 6 months of life
* Suspected or proven metabolic diseases
* No parental/guardian consent

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with congenital heart disease requiring a first intervention within the first 6 months of life
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical neurological development measured with Bayley Scale of Infant Development | 9 months, 24 months
  Rate of abnormal clinical neurodevelopment measured with the Bayley Scale of Infant Development (BSID-III): range 50-150, mean 100, SD 15
Brain MRI structural brain abnormalities | +- 1 week postoperative
  Incidence of patients with normal brain development vs rate of bleeding/stroke visualized on brain MRI Differences in total brain volume and cerebellar volume in patients with congenital heart disease

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No